CLINICAL TRIAL: NCT02188862
Title: Genome-wide Association Study of Susceptibility to Rheumatic Heart Disease in Fiji and New Caledonia
Brief Title: Genetic Susceptibility to Rheumatic Heart Disease in the Pacific Region
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Ministry of Health, Fiji (Other Government); Fiji National University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut Necker Enfants Malades (Other); Centre Hospitalier Territorial de Nouvelle-Calédonie (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Other Study IDs: PACIFICRHDGEN
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatic Heart Disease; Mitral Stenosis
Keywords: Rheumatic heart disease; Acute rheumatic fever; Group A streptococcal disease; Streptococcus pyogenes; Genetics; Oceania
MeSH Terms: conditions — Rheumatic Heart Disease; Mitral Valve Stenosis; Rheumatic Fever; Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood collected from all participants for extraction of DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatic heart disease cases: Patients with rheumatic heart disease as defined in the case criteria
- Population controls: Individuals from the general population divided into new controls (recruited specifically for this study) and existing controls (recruited to previous population genetics studies in the region)

SUMMARY:
The purpose of this study is to investigate whether there are genetic differences between patients with rheumatic heart disease and members of the general population.

DETAILED DESCRIPTION:
The investigators will micro-array genotype approximately 300,000 single nucleotide polymorphisms (SNP) using DNA samples from patients with rheumatic heart disease (cases) from New Caledonia and Fiji, and members of the general population (controls) from New Caledonia, Vanuatu and Fiji. The investigators will perform standard quality control checks on the SNP data using measures such as call rate, heterozygosity, duplication and relatedness, and exclude variants on the basis of deviation from Hardy-Weinberg equilibrium and minor allele frequency. We will also impute variants not present on the micro-array with reference to the latest release of 1000 Genomes data and whole-genome sequence data from sixty Melanesian individuals from New Caledonia from the phenotypic extremes in this study.

The investigators will conduct a discovery analysis in using a genome-wide association study approach focusing on Oceanic cases and controls from the Francophone nations of New Caledonia and Vanuatu. This analysis will be corrected for bias due to population stratification using the Linear Mixed Model (LMM) and consider additive, dominant and recessive genetic models. The investigators will then perform LMM association testing for variants with P-value in the discovery analysis less than 1x10^-5 in Oceanic cases and controls from Fiji and combine the association statistics by fixed-effects meta-analysis. The investigators will consider variants with significant effects in the same direction in discovery and replication analyses with combined P-value less than 1x10^-8 to have replicated. Unless there is clear evidence that associated variants are specific to Oceanic populations, further replication analyses for associated variants in cases and controls of Indian Descent from Fiji, as well as individuals of other and admixed ethnicities from both Fiji and New Caledonia.

Recruitment completed in December 2013. After receipt of funding from the British Heart Foundation, genotyping and analysis will begin in July 2014.

ELIGIBILITY:
1. Cases

   1. Inclusion Criteria:

      * Diagnosis of rheumatic heart disease based on one of:

        * World Heart Federation definite echocardiographic criteria
        * World Heart Federation borderline echocardiographic criteria and history of acute rheumatic fever
        * Mitral stenosis with valve area less than 2.0 cm2
        * Previous surgery for rheumatic heart disease
   2. Exclusion Criteria:

      * Age less than five years
      * Inability to give consent
2. New Controls

   1. Inclusion criteria:

      * Healthy individual living in a community where cases were identified
   2. Exclusion Criteria:

      * Past medical history or systems suggestive of rheumatic heart disease, acute rheumatic fever or other valvular heart disease
      * Age less than five years
      * Inability to give consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases:
  * Prevalent and incident cases of rheumatic heart disease ascertained from disease registers, primary care clinics and hospital services.
  New Controls:
  * Individuals volunteering from communities where cases were identified.
  Existing Controls:
  * Individuals from this region who have previously been recruited to population genetics research studies.
Sampling Method: Non-Probability Sample
Enrollment: 2372 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rheumatic heart disease diagnosis | At enrolment
  Diagnosis of rheumatic heart disease as layout in enrolment criteria for cases.

SECONDARY OUTCOMES:
Mitral stenosis diagnosis | At enrolment
  History or echocardiographic diagnosis of mitral stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Tom Parks, MRCP DTM&H, Principal Investigator — University of Oxford; Mariana Mirabel, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Andrew C Steer, FRACP PhD, Principal Investigator — University of Melbourne; Adrian VS Hill, DPhil DM, Study Chair — University of Oxford
Locations (3):
- Colonial War Memorial Hospital, Suva, Fiji
- Centre Hospitalier Territorial de Nouvelle Caledonie, Noumea, New Caledonia
- Wellcome Trust Centre for Human Genetics, University of Oxford, Oxford, United Kingdom

REFERENCES:
- See also: Link to study documents and protocols — http://users.ox.ac.uk/~clme1250/rhd_consortium/pacific.html